CLINICAL TRIAL: NCT05884398
Title: A Phase 3, Open-label, Randomized, Prospective Study of Apalutamide With Continued Versus Intermittent Androgen-Deprivation Therapy (ADT) Following PSA Response in Participants With Metastatic Castration-Sensitive Prostate Cancer (mCSPC)
Brief Title: A Study of an Intermittent ADT Approach With Apalutamide Monotherapy in Participants With mCSPC
Acronym: LIBERTAS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109327; 56021927PCR3020 (Other: Janssen Research & Development, LLC); 2022-502686-24-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castrate-sensitive Prostate Cancer
MeSH Terms: interventions — apalutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Intermittent ADT Group) (Experimental): Participants with PSA level <0.2 ng/mL after 6 months of treatment with Apalutamide and ADT during initial treatment phase, will enter main treatment phase and treated with apalutamide with intermittent ADT per protocol or followed up for at least 18 months from Day 1 of Cycle 7 (each cycle 28 days) and followed up for up to a maximum of 2 years after the main treatment phase, or until death, withdrawal of consent, loss to follow-up, early termination of the study by the sponsor for any reason, whichever occurs first.
  Interventions: Drug: Apalutamide; Drug: Androgen-deprivation Therapy (ADT)
- Arm B (Continuous ADT Group) (Active Comparator): Participants with PSA level <0.2 ng/mL after 6 months of treatment with Apalutamide and ADT during initial treatment phase, will enter main treatment phase and continue to receive apalutamide plus ADT or followed up for at least 18 months from Day 1 of Cycle 7 (each cycle 28 days) and followed up for up to a maximum of 2 years after the main treatment phase, or until death, withdrawal of consent, loss to follow-up, early termination of the study by the sponsor for any reason, whichever occurs first.
  Interventions: Drug: Apalutamide; Drug: Androgen-deprivation Therapy (ADT)

INTERVENTIONS:
Drug: Apalutamide — Apalutamide will be administered orally from Day 1 of Cycle 1 till 6 months in initial treatment phase and then in main treatment phase from Day 1 of Cycle 7 up to at least 18 months.
Drug: Androgen-deprivation Therapy (ADT) — The choice of ADT will be at discretion of the Investigator. Dosing (dose and frequency of administration) will be consistent with the prescribing information.

SUMMARY:
The purpose of the study is to determine if the intermittent use of androgen-deprivation therapy (ADT) in participants with metastatic castrate-sensitive prostate cancer (mCSPC) who reached a prostate-specific antigen (PSA) level < 0.2 nanograms/millilitres (ng/mL) after 6 months of treatment with apalutamide and ADT combination therapy provides non-inferior radiographic progression-free survival (rPFS) and a reduced burden of hot flashes measured as 18-month percent change in severity adjusted hot flash score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer prior to screening with histologically or cytologically confirmed adenocarcinoma of the prostate
* For participants not undergoing Gender-affirming care: Metastatic prostate cancer disease documented by conventional imaging (example, computed tomography [CT], magnetic resonance imaging [MRI], or bone scan) and/or next-generation imaging [NGI] demonstrating greater than or equal (>=) 2 distinct extraprostatic sites of metastasis
* For participants undergoing Gender-affirming care: No evidence of metastasis by either conventional imaging (example, CT, MRI, or bone scan) and/or NGI is also acceptable
* For participants not undergoing gender-affirming care: testosterone levels > 50 (ng/dL) nanograms per deciliter at screening, except for those who may have received ADT prior to screening. Participants are allowed to have received up to 3 months of (ADT) androgen-deprivation therapy prior to enrollment
* For participants undergoing Gender-affirming care: There is no testosterone level requirement for inclusion
* Have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1. Participants with ECOG PS 2 or 3 are eligible for the study if the ECOG PS score is related to stable physical limitations (example, wheelchair-bound due to prior spinal cord injury) and not related to prostate cancer or associated therapy
* A participant must agree not to plan to conceive a child while enrolled in this study or within 3 months after the last dose of study treatment
* Must be able to take whole apalutamide tablets by swallowing alone or with another vehicle (example, applesauce)
* Assigned male at birth, inclusive of all gender identities

Exclusion Criteria:

* History of seizure or known condition that has been determined to significantly predispose to seizure per investigator
* Pelvic lymph nodes as only site of metastasis
* Known allergies, hypersensitivity, or intolerance to excipients of apalutamide
* Any of the following within 6 months prior to screening: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, uncontrolled hypertension, clinically significant arterial or venous thromboembolic events
* Gastrointestinal disorder affecting absorption
* Participants who have undergone a bilateral orchiectomy with the exception of participants who completed this as part of their gender-affirming care or a result of a variation in physical sex development

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male assigned at birth, inclusive of all gender identities.
Enrollment: 420 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2028-10-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With 18-Months Radiographic Progression-free Survival (rPFS) | From randomization (Day 1 of Cycle 7) up to 18 months
  rPFS is defined as the duration from the date of randomization to the date of first documentation of confirmed radiographic progressive disease or death due to any cause, whichever occurs first. rPFS will be assessed by investigators using conventional imaging (computed tomography [CT]/magnetic resonance imaging [MRI] and 99mTc bone scans).
Percent Change From Randomization in Severity of Adjusted Hot Flash Score at 18 Months | From randomization (Day 1 of Cycle 7) up to 18 months
  Severity adjusted hot flash score will be calculated from the hot flash diary which will be daily filled by the participants.

SECONDARY OUTCOMES:
Mean Percentage Changes From Randomization in Severity Adjusted Hot Flash Score and Hot Flash Frequency | From randomization (Day 1 of Cycle 7), up to 5 years
  Severity adjusted hot flash score and hot flash frequency will be calculated from the hot flash diary which will be daily filled by the participants.
Second Progression-free Survival (PFS2) | From randomization (Day 1 of Cycle 7) up to 5 years
  PFS2 is defined as the duration from the date of randomization to the first occurrence of investigator-determined disease progression on the first subsequent therapy after study drug discontinuation or death, whichever occurs first.
Overall Survival (OS) | From randomization (Day 1 of Cycle 7) up to 5 years
  Overall survival time is defined as the duration from the date of randomization to the date of death from any cause.
Prostate Cancer-specific Survival | From randomization (Day 1 Cycle 7) up to 5 years
  Prostate cancer-specific survival is defined as the duration from the date of randomization to the date of death from prostate cancer-specific cause.
Serum Prostate Specific Antigen (PSA) Evaluations | From randomization (Day 1 of Cycle 7) up to 5 years
  Serum PSA evaluations will be measured according to Prostate Cancer Working Group 3 (PCWG3) criteria.
Duration of Time on Androgen-deprivation Therapy (ADT) | From randomization (Day 1 of Cycle 7) up to 5 years
  Duration of time on ADT will be reported for all participants.
Time to First ADT Restart | From randomization (Day 1 of Cycle 7) up to 5 years
  Time to first ADT restart will be reported.
Duration of Time with Testosterone Level Less than (<) 50 nanograms per millilitre (ng/mL) | From randomization (Day 1 of Cycle 7) up to 5 years
  Duration of time with testosterone level <50 ng/mL will be reported.
Time to Recovery of Testosterone >50 nanogram per decilitre (ng/dL) | From randomization (Day 1 of Cycle 7) up to 5 years
  The testosterone recovery, defined as a serum testosterone >50 ng/dL will be analyzed.
Time to Recovery of Testosterone Greater Than or Equal (>=) Screening Testosterone Level | From randomization (Day 1 of Cycle 7) up to 5 years
  Time to recovery of testosterone >= screening testosterone level will be reported.
Time to Testosterone Recovery to Normal Range (>270 ng/dL) | From randomization (Day 1 of Cycle 7) up to 5 years
  Time to serum testosterone recovery to normal range (>270 ng/dL) will be reported.
Time to Metastatic Castration-resistant Prostate Cancer (mCRPC) | From randomization (Day 1 of Cycle 7) up to 5 years
  Time to mCRPC will be reported.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Initial Treatment Phase: From Day 1 of Cycle 1 (each cycle 28 days) up to end of Cycle 6 (6 month); Main Treatment Phase: Day 1 of Cycle 7 up to end of study (up to 5 years)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, or is an important medical event.
Number of Participants with Abnormal Clinical Laboratory Parameters | From Cycle 1 Day 1 up to 5 years
  Number of participants with abnormal clinical laboratory parameters (hematology, clinical chemistry) will be reported.
Number of Participants with Abnormal Vital Sign Parameters | From Cycle 1 Day 1 up to 5 years
  Number of participants with abnormal vital sign parameters (temperature, pulse/heart rate, respiratory rate, and blood pressure) will be reported.
Number of Participants with Abnormal Physical Examination Parameters | From Cycle 1 Day 1 up to 5 years
  Number of Participants with Abnormal physical examination parameters will be reported.
Hot Flash Related Daily Interference Score (HFRDIS) | Up to 5 years
  The HFRDIS is a 10-item scale assessing how much hot flashes interfered with various aspects of a participant's daily life. All items are rated on a 0-10 numerical rating scale with 0 anchored as "Do Not Interfere" and 10 as "Completely Interfere." A total score is computed by summing items. Higher scores indicate higher interference due to hot flashes and thus, greater impact on quality of life.
Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | Baseline up to 5 years
  The EORTC-QLQ-C30 (Version 3), is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. The recall period for most items is the past week. EORTC-QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status/quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire -Prostate Cancer Module (EORTC-PR25) Questionnaire | Baseline up to 5 years
  The EORTC-PR25 questionnaire is a supplement to the EORTC-QLQ-C30 questionnaire and is designed to assess symptoms related to prostate cancer, its treatment, and aspects of life related to this type of cancer.
Change From Baseline in European Organization for the Research and Treatment of Cancer (EORTC) Customized Study Form | Baseline up to 5 years
  EORTC customized study form will include 3 questions that are not included on the QLQ-30 or PR25 forms. The items assess rash, side effect burden, and dry mouth.
Change From Baseline in Patient-Reported Outcomes Measurement Information System Cognitive Function (PROMIS-Cog) Questionnaire | Baseline up to 5 years
  The PROMIS-Cog is a self-administered fixed-length questionnaire of 8 items from the PROMIS item bank relating to cognitive function. The raw domain scores are converted to standardized T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate better cognitive functioning.
Change From Baseline in Memorial Anxiety Scale for Prostate Cancer (MAX-PC) Questionnaire | Baseline up to 5 years
  The MAX-PC is a patient-reported questionnaire measuring prostate cancer specific anxiety. It consists of 18 items in 3 domains: It includes 11 items regarding prostate cancer anxiety, scored 0-33; 3 items regarding prostate-specific Antigen Anxiety, scored 0-9; and 4 items regarding fear of recurrence, scored 0-12. Total score ranges from 0-54 with higher scores indicating greater anxiety.
Change From Baseline in Patient Health Questionnaire (PHQ-9) Questionnaire | Baseline up to 5 years
  The PHQ-9 is self-administered, 9-item questionnaire measuring symptoms of depression. The recall period for all items is the past 2 weeks. The items include diminished interest or pleasure, depressed mood, insomnia/hypersomnia, fatigue or loss of energy, weight loss or weight gain/appetite loss or appetite gain, feelings of worthlessness, diminished concentration/indecisiveness, psychomotor agitation/retardation, and thoughts of death/suicide. Higher scores indicate more severe depressive symptoms.
Change From Baseline in Patient Global Impression of Severity scale (PGIS) Questionnaire | Baseline up to 5 years
  The PGIS is a self-administered, single item questionnaire measuring patients' impression of disease severity. Participants will be asked to rate their disease severity over the past 7 days using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe. Higher scores indicate greater severity of fatigue.
Change From Baseline in Patient Global Impression of Change (PGIC) Questionnaire | Baseline up to 5 years
  The PGIC is self-administered, single-item questionnaire measuring patients' impression of change in disease symptoms. Participants will be asked to rate their current symptoms as compared to when they started the study, using the following 7-point scale: 1 = Much better, 2 = Moderately better, 3 = A little better, 4 = No change, 5 = A little worse, 6 = Moderately worse, and 7 = Much worse. A higher PGIC score indicates greater worsening of symptoms.
Time to Recovery From Baseline as Assessed by EORTC-QLQ-C30 | Baseline up to 5 years
  Time to recovery from baseline as assessed by EORTC-QLQ-C30 will be reported. The EORTC-QLQ-C30 (Version 3), is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. The recall period for most items is the past week. EORTC-QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status/quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Time to Recovery From Baseline as Assessed by EORTC-PR25 | Baseline up to 5 years
  Time to recovery from baseline as assessed by EORTC-PR25 will be reported. The EORTC-PR25 questionnaire is a supplement to the EORTC-QLQ-C30 questionnaire and is designed to assess symptoms related to prostate cancer, its treatment, and aspects of life related to this type of cancer.
Time to Recovery From Baseline as Assessed by EORTC Customized Study Form | Baseline up to 5 years
  Time to recovery from baseline as assessed by EORTC customized study form will be reported. EORTC customized study form will include 3 questions that are not included on the QLQ-30 or PR25 forms. The items assess rash, side effect burden, and dry mouth.
Time to Recovery From Baseline as Assessed by MAX-PC | Baseline up to 5 years
  Time to recovery from baseline as assessed by MAX-PC will be reported. The MAX-PC is a patient-reported questionnaire measuring prostate cancer specific anxiety. It consists of 18 items in 3 domains: It includes 11 items regarding prostate cancer anxiety, scored 0-33; 3 items regarding prostate-specific Antigen Anxiety, scored 0-9; and 4 items regarding fear of recurrence, scored 0-12. Total score ranges from 0-54 with higher scores indicating greater anxiety.
Time to Recovery From Baseline as Assessed by PHQ-9 | Baseline up to 5 years
  Time to recovery from baseline as assessed by PHQ-9 will be reported. The PHQ-9 is self-administered, 9-item questionnaire measuring symptoms of depression. The recall period for all items is the past 2 weeks. The items include diminished interest or pleasure, depressed mood, insomnia/hypersomnia, fatigue or loss of energy, weight loss or weight gain/appetite loss or appetite gain, feelings of worthlessness, diminished concentration/indecisiveness, psychomotor agitation/retardation, and thoughts of death/suicide. Higher scores indicate more severe depressive symptoms.
Time to Recovery From Baseline as Assessed by PGIS | Baseline up to 5 years
  Time to recovery from baseline as assessed by PGIS will be reported. The PGIS is a self-administered, single item questionnaire measuring patients' impression of disease severity. Participants will be asked to rate their disease severity over the past 7 days using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe. Higher scores indicate greater severity of fatigue.
Time to Recovery From Baseline as Assessed by PGIC | Baseline up to 5 years
  Time to recovery from baseline as assessed by PGIC will be reported. The PGIC is self-administered, single-item questionnaire measuring patients' impression of change in disease symptoms. Participants will be asked to rate their current symptoms as compared to when they started the study, using the following 7-point scale: 1 = Much better, 2 = Moderately better, 3 = A little better, 4 = No change, 5 = A little worse, 6 = Moderately worse, and 7 = Much worse. A higher PGIC score indicates greater worsening of symptoms.
Time to Recovery From Baseline as Assessed by PROMIS-Cog | Baseline up to 5 years
  Time to recovery from baseline as assessed by PROMIS-Cog will be reported. The PROMIS-Cog is a self-administered fixed-length questionnaire of 8 items from the PROMIS item bank relating to cognitive function. The raw domain scores are converted to standardized T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate better cognitive functioning.
Time to Deterioration in EORTC-QLQ-C30 Over Time | Up to 5 years
  Time to deterioration in EORTC-QLQ-C30 over time will be reported. The EORTC-QLQ-C30 (Version 3), is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. The recall period for most items is the past week. EORTC-QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status/quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Time to Deterioration in EORTC-PR25 Over Time | Up to 5 years
  Time to deterioration in EORTC-PR25 over time will be reported. The EORTC-PR25 questionnaire is a supplement to the EORTC-QLQ-C30 questionnaire and is designed to assess symptoms related to prostate cancer, its treatment, and aspects of life related to this type of cancer.
Time to Deterioration in EORTC Customized Study Form Over Time | Up to 5 years
  Time to deterioration in EORTC Customized Study Form over time will be reported. EORTC customized study form will include 3 questions that are not included on the QLQ-30 or PR25 forms. The items assess rash, side effect burden, and dry mouth.
Time to Deterioration as per PROMIS-Cog Questionnaire Over Time | Up to 5 years
  Time to deterioration as per PROMIS-Cog questionnaire over time will be reported. The PROMIS-Cog is a self-administered fixed-length questionnaire of 8 items from the PROMIS item bank relating to cognitive function. The raw domain scores are converted to standardized T-scores with a mean of 50 and a standard deviation of 10. Higher scores indicate better cognitive functioning.
Time to Deterioration in MAX-PC Questionnaire Over Time | Up to 5 years
  Time to deterioration in MAX-PC questionnaire over time will be reported. The MAX-PC is a patient-reported questionnaire measuring prostate cancer specific anxiety. It consists of 18 items in 3 domains: It includes 11 items regarding prostate cancer anxiety, scored 0-33; 3 items regarding prostate-specific Antigen Anxiety, scored 0-9; and 4 items regarding fear of recurrence, scored 0-12. Total score ranges from 0-54 with higher scores indicating greater anxiety.
Time to Deterioration as per PHQ-9 Questionnaire Over Time | Up to 5 years
  Time to deterioration as per PHQ-9 questionnaire over time will be reported. The PHQ-9 is self-administered, 9-item questionnaire measuring symptoms of depression. The recall period for all items is the past 2 weeks. The items include diminished interest or pleasure, depressed mood, insomnia/hypersomnia, fatigue or loss of energy, weight loss or weight gain/appetite loss or appetite gain, feelings of worthlessness, diminished concentration/indecisiveness, psychomotor agitation/retardation, and thoughts of death/suicide. Higher scores indicate more severe depressive symptoms.
Time to Deterioration in PGIS Questionnaire Over Time | Up to 5 years
  Time to deterioration as per PGIS questionnaire over time will be reported. The PGIS is a self-administered, single item questionnaire measuring patients' impression of disease severity. Participants will be asked to rate their disease severity over the past 7 days using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe. Higher scores indicate greater severity of fatigue.
Time to Deterioration as per PGIC Questionnaire Over Time | Up to 5 years
  Time to Deterioration as per PGIC questionnaire over time will be reported. The PGIC is self-administered, single-item questionnaire measuring patients' impression of change in disease symptoms. Participants will be asked to rate their current symptoms as compared to when they started the study, using the following 7-point scale: 1 = Much better, 2 = Moderately better, 3 = A little better, 4 = No change, 5 = A little worse, 6 = Moderately worse, and 7 = Much worse. A higher PGIC score indicates greater worsening of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (93):
- United States (46):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Arizona Urology Specialists, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Urology Associates of Central California, Fresno, California
  - VA Medical Center, San Francisco, California
  - Sansum Clinic Pharm, Santa Barbara, California
  - Colorado Clinical Research, Lakewood, Colorado
  - Advanced Urology Institute, Daytona Beach, Florida
  - Associated Urological Specialists LLC, Chicago Ridge, Illinois
  - Advanced Urology Associates, Joliet, Illinois
  - Urology of Indiana, Greenwood, Indiana
  - First Urology, PSC, Jeffersonville, Indiana
  - Maryland Oncology Hematology P A, Silver Spring, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - MSKCC Basking Ridge, Basking Ridge, New Jersey
  - MSKCC Monmouth, Middletown, New Jersey
  - MSKCC Bergen, Montvale, New Jersey
  - MSKCC Commack, Commack, New York
  - MSKCC Westchester, Harrison, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Associated Medical Professionals, Syracuse, New York
  - MSKCC Nassau Regional Cancer Center, Uniondale, New York
  - TriState Urologic Services PSC Inc. DBA The Urology Group, Cincinnati, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Helios Clinical Research, LLC, Middleburg Heights, Ohio
  - Northwest Cancer Specialists PC, Tigard, Oregon
  - Centers for Advanced Urology LLC d b a MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - VA Pittsburgh, Pittsburgh, Pennsylvania
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Texas Oncology P A, Austin, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - Texas Oncology P A, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology P A, Houston, Texas
  - Houston Metro Urology, Houston, Texas
  - Texas Oncology San Antonio Northeast, San Antonio, Texas
  - Texas Oncology P A, Wichita Falls, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Urology Of Virginia, Pllc, Virginia Beach, Virginia
- Australia (3):
  - Macquarie University Hospital, Macquarie University
  - Peter MacCallum Cancer Centre, Melbourne
  - Mater Misericordiae Hospital, South Brisbane
- Brazil (7):
  - Fundacao Pio XII, Barretos
  - Hospital das Clínicas - Universidade Federal de Minas Gerais, Belo Horizonte
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino, Salvador
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Fundacao Faculdade de Medicina Instituto do Cancer do Estado de Sao Paulo, São Paulo
- Canada (5):
  - Southern Alberta Institute of Urology / Prostate Cancer Centre, Calgary, Alberta
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHU de Quebec Universite Laval Hopital de l Enfant Jesus, Québec, Quebec
- China (10):
  - Peking University First Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China School of Medicine/West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - Nanfang Hospital of Southern Medical Hospital, Guangzhou
  - Shandong Provincial Hospital, Jinan
  - Ningbo First Hospital, Ningbo
  - Shengjing Hospital Of China Medical University, Shenyang
  - TongJi Hospital of TongJi Medical College of Huazhong University of Science & Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Hopital Cochin, Paris
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Gustave Roussy, Villejuif
- Germany (8):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Universitaetsklinikum Koelnt, Cologne
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Klinikum rechts der Isar - der Technischen Universität München, München
  - Studienpraxis Urologie Nurtingen, Nürtingen
  - Universitatsklinikum Wurzburg, Würzburg
- Mexico (4):
  - SCIENTIA Investigacion Clinica SC, Chihuahua City
  - Consultorio de Especialidad en Urologia Privado, Durango
  - Medical Care & Research SA de CV, Mérida
  - Cuidados Oncologicos, Querétaro
- Poland (5):
  - Centrum Onkologii im Prof F Lukaszczyka, Bydgoszcz
  - Szpital Wojewodzki im Mikolaja Kopernika w Koszalinie, Koszalin
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Szpital Grochowski Im Dr Med Rafala Masztaka Sp Z O O, Warsaw
  - Polimed Specjalistyczna Przychodnia Lekarska Wieslaw Grazyna Tupikowski Bednarek Tupikowska S C, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency